CLINICAL TRIAL: NCT06151548
Title: Effect of Krill Oil Supplementation on Red Blood Cell Physiology Against Changes in Markers of Iron Metabolism.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: jcichonwozniakZWKF
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-11

CONDITIONS: Red Blood Cell Disorder; Oxidative Stress; Iron Metabolism Disorders
MeSH Terms: conditions — Iron Metabolism Disorders | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: All competitors will be randomly divided into two groups (double-blind):
  A. supplemented (n = 15), who will receive three times a day one capsule of a supplement called THYROX (Atlantic krill oil).
  B. control (n = 15) receiving placebo. The supplementation period will be six weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: the Polish Youth Rowing Team
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supplemented (Experimental): (n = 15), who will receive four times a day one capsule of a supplement called THYROX (Atlantic krill oil). The daily content of krill oil is 2000 mg, including omega-3 fatty acids 350 mg, EPA - 240 mg, DHA - 110 mg, phospholipids - 800 mg, astaxanthin 200 mg.
  The supplementation period will be six weeks.
  Interventions: Drug: THYROX (Atlantic krill oil).
- control (Experimental): receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THYROX (Atlantic krill oil). — The daily content of krill oil is 2000 mg, including omega-3 fatty acids 350 mg, EPA - 240 mg, DHA - 110 mg, phospholipids - 800 mg, astaxanthin 200 mg.
  Arms: supplemented
Drug: Placebo — The control capsules will be made of olive oil of equal size and color.
  Arms: control

SUMMARY:
Research group: the research will be conducted in a homogeneous group of professional rowers (N=30), all competitors qualified for the Polish Youth Rowing Team:

* aged 18 - 24, because the age group must be homogeneous,
* the size of the group is about thirty people, which in the case of a homogeneous group will enable statistical analyzes to be conducted.

Rowing performance test: at the beginning and at the end of the training camp, participants will perform a test on a rowing ergometer (Concept II, USA), each subject will have to cover a distance of 2000 m in the shortest possible time, which is the distance starting in rowing competitions. The results of both tests will be considered in the selection for the championship team; therefore, athletes will be well motivated to perform both tests with maximum effort.

The investigators set a research hypothesis that supplementation with krill oil may have a beneficial effect on athletes by limiting lipid peroxidation and inhibiting ferroptosis which in consequence may lead to red blood cell membrane protection.

DETAILED DESCRIPTION:
All competitors will be randomly divided into two groups (double-blind):

A. supplemented (n = 15), who will receive four times a day one capsule of a supplement called THYROX (Atlantic krill oil). The daily content of krill oil is 2000 mg, including omega-3 fatty acids 350 mg, EPA - 240 mg, DHA - 110 mg, phospholipids - 800 mg, astaxanthin 200 mg.The supplementation period will be six weeks.

B. control (n = 15) receiving placebo. MLB Biotrade Sp. z o. o., Poznan, Poland will produce all oil krill supplements and placebo.

Measurement: All determined parameters will be measured with the available equipment in the ZWKF laboratory in Gorzów Wielkopolski and using commercial assay kits. Measurements will be performed by the project contractors.

1. Polyethylene tubes (2.7ml) containing dipotassium ethylenediaminetetraacetic acid (EDTAK2) anticoagulant will be used for the following tests:

   1. complete blood count (18 parameters) determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland). White blood cell indices: WBC (white blood cells), LYM (lymphocytes as a percentage), LYM (lymphocytes), MON (monocytes as a percentage), MON (monocytes), GRA (granulocytes as a percentage), GRA (granulocytes). Red blood cell indices: RBC (Red Blood Cells), HGB (Hemoglobin), HCT (Hematocrit), MCV (Mean Corpuscular Volume), MCH (Mean Corpuscular Hemoglobin), MCHC (Mean Corpuscular Hemoglobin Concentration), RDW (Red Blood cells Distribution Width). Platelet indices: PLT (Platelet), MPV (Mean Platelet Volume), PDW (Platelet Distribution Width), PCT (Thrombocrit).
   2. a manual blood smear will be made by placing a drop of blood on a slide and then spreading it with a uniform motion. After drying, it will be colored by the May Grunwald-Giemsa method according to the procedure. The stained and fixed smear after drying will be viewed under a microscope for quantitative and qualitative assessment.
   3. reticulocyte count will be performed by incubating the collected blood with reticulocyte dye in the proportion specified by the manufacturer. Next, a smear will be made, and after drying, the number of cells will be counted.
2. Polyethylene clotting activator tubes (9 ml) will be centrifuged to separate the morphotic elements from the serum using a centrifuge (3000 rpm for 10 min). The serum will be pipetted into several Eppendorf tubes, which will then be frozen (temp. -80 °C). All the following biochemical parameters will be determined from the extracted serum:

   1. using the ELISA method by the test manufacturer's instructions. The designations include the flowing parameters:

      * markers of oxidative stress: 4-Hydroxynonenal (4-HNE), Total Antioxidant Capacity (TAC), Heme oxygenase 1 (HO-1) and 8-Isoprostane.
      * iron status parameters: hepcidin, soluble transferrin receptor, ferritin, erythroferrone, lactoferrin
      * indicators of muscle damage: myoglobin.
   2. the iron and Total Iron Binding Capacity (TIBC) levels (Unsaturated Iron Binding Capacity (UIBC) will be calculated from the formula: UIBC = TIBC-iron in serum) will be determined using the colorimetric method on the SPECTROstar Nano reader.
3. The lactate (La) concentration will be determined from the capillary blood immediately after collection using a commercially available kit (Dr. Lange, Germany).

ELIGIBILITY:
Inclusion Criteria:

* training experience a minimum of five years
* minimum training time per week 240 minutes
* all competitors qualified for the Polish Youth Rowing Team

Exclusion Criteria:

* health problems,
* antibiotic therapy,
* taking other supplements during the study period or a month earlier

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-23 (Estimated); Primary Completion 2024-06-24 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
complete blood count | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  (18 parameters) determined on the MYTHIC 18 hematology analyzer (Orphee Medical, Geneva, Switzerland). White blood cell indices: WBC (white blood cells), LYM (lymphocytes as a percentage), LYM (lymphocytes), MON (monocytes as a percentage), MON (monocytes), GRA (granulocytes as a percentage), GRA (granulocytes). Red blood cell indices: RBC (Red Blood Cells), HGB (Hemoglobin), HCT (Hematocrit), MCV (Mean Corpuscular Volume), MCH (Mean Corpuscular Hemoglobin), MCHC (Mean Corpuscular Hemoglobin Concentration), RDW (Red Blood cells Distribution Width). Platelet indices: PLT (Platelet), MPV (Mean Platelet Volume), PDW (Platelet Distribution Width), PCT (Thrombocrit).
a manual blood smear | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  will be made by placing a drop of blood on a slide and then spreading it with a uniform motion. After drying, it will be colored by the May Grunwald-Giemsa method according to the procedure. The stained and fixed smear after drying will be viewed under a microscope for quantitative and qualitative assessment.
reticulocyte count | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  will be performed by incubating the collected blood with reticulocyte dye in the proportion specified by the manufacturer. Next, a smear will be made, and after drying, the number of cells will be counted.
markers of oxidative stress | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  4-Hydroxynonenal (4-HNE), Total Antioxidant Capacity (TAC), Heme oxygenase 1 (HO-1)and 8-Isoprostane. ELISA method by the test manufacturer's instructions
iron status parameters | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  hepcidin, soluble transferrin receptor, ferritin erythroferrone and lactoferrin. ELISA method by the test manufacturer's instructions
indicators of muscle damage | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  mioglobin. ELISA method by the test manufacturer's instructions
The iron and TIBC | Blood samples will be taken from the cubital vein at three-time points: before each stress test (after overnight fasting), one minute after the end of the test, and after a 3-hour recovery period.
  the iron and Total Iron Binding Capacity (TIBC) levels (Unsaturated Iron Binding Capacity (UIBC) will be calculated from the formula: UIBC = TIBC-iron in serum) will be determined using the colorimetric method on the SPECTROstar Nano reader.

CONTACTS AND LOCATIONS:
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No